CLINICAL TRIAL: NCT02743182
Title: HBsAg Loss Adding Pegylated Interferon Alfa-2a in HBeAg-negative Patients Treated With Nucleos(t)Ide Analogues.
Brief Title: HBsAg Loss Adding Pegylated Interferon in HBeAg-negative Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: José Antonio Carrion (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor-Investigator, José Antonio Carrion, Dr., Parc de Salut Mar
Organization: Parc de Salut Mar (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: QUANTI-B
Record Dates: First submitted 2016-04-12; First posted 2016-04-19 (Estimated); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Chronic Hepatitis B (HBeAg-negative)
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pegylated interferon alfa-2a (Active Comparator): adding Pegylated interferon alfa-2a (180 microgs /week during 48 weeks) in HBeAg-negative patients receiving nucleos(t)ide analogues
  Interventions: Drug: Pegylated interferon alfa-2a
- Control (No Intervention): HBeAg-negative patients receiving nucleos(t)ide analogues

INTERVENTIONS:
Drug: Pegylated interferon alfa-2a
  Arms: Pegylated interferon alfa-2a

SUMMARY:
Chronic hepatitis B (CHB) affects more than 350 million people worldwide. The most common form in Europe is CHB HBeAg-negative. Antiviral treatment of CHB HBeAg-negative patients includes chronic administration of nucleos(t)ide analogues (NUC) or pegylated interferon (PegIFN) during 12 months. Typically, PegIFN allows immune control of CHB and antigen "s" (HBsAg) loss in around 4% of patients compared to less than 0,1% using NUC. Recently, it has been described that HBsAg quantification (HBsAg-q) is useful to identify patients with high probability to lose HBsAg during follow-up. In addition, a proof-of-concept study with nine HBeAg-negative patients receiving NUC showed that adding PegIFN (16 weeks) achieved HBsAg loss in one patient (11%). The aim of our study is to evaluate the efficacy and safety adding PegIFN (48 weeks) in treated HBeAg-negative patients with NUC.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis B (HBeAg-negative)
* Signed inform consent
* Aged > 18

Exclusion Criteria:

* Contraindications for Pegylated interferon (cirrhosis, pregnancy, others)
* Previous treatment with interferon or Pegylated interferon
* Previous HBsAg loss
* Treatment duration with Nucleos(t)ide analogues less than 2 years
* Poor adherence to Nucleos(t)ide analogues

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2015-01; Primary Completion 2018-10 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Number of patients with HBsAg loss | 1 year after treatment completion
  HBsAg will be evaluated one year after treatment completion (96 weeks). Efficacy will be calculated as a proportion (rate of patients with HBsAg loss/treated patients)